CLINICAL TRIAL: NCT02838342
Title: Pharmaco-immunological Study of Interferon-alpha and Metronomic Cyclophosphamide Association in Neuroendocrine Tumors
Acronym: EPICentro
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: API/2015/61
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Interferon-alpha

ARMS (1):
- Metronomic cyclophosphamide and interferon-alpha (Experimental)
  Interventions: Drug: Metronomic cyclophosphamide; Drug: Interferon-alpha

INTERVENTIONS:
Drug: Metronomic cyclophosphamide — 50 mg oral tablet, one tablet per day, every day for 6 months; abort if progression or intolerance
  Other Names: CMC
Drug: Interferon-alpha — 3 months of treatment from the 4th cycle metronomic cyclophosphamide : subcutaneous injection, initial dose of 3 MIU three times a week. The dose may be adjusted as tolerated to achieve a T cell counts greater than 500 / mm3
  Other Names: IFN-alpha

SUMMARY:
This study will evaluate the potential immunomodulatory synergy of the association of metronomic cyclophosphamide (CMC) and interferon-alpha (IFN-alpha).

ELIGIBILITY:
Inclusion Criteria:

* performance status ECOG-WHO ≤ 1
* histologically proved neuroendocrine tumor with Ki67 < or = 10%, metastatic or locally advanced without surgery possibility
* at least one measurable lesion based on RECIST criteria version 1.1
* signed written informed consent

Exclusion Criteria:

* previous treatment with interferon or cyclophosphamide
* treatment by immunosuppressive drugs
* diabetes complicated by coronary artery disease or vasculopathy
* severe respiratory failure, chronic respiratory failure, COPD
* history of severe heart failure
* severe renal or hepatic impairment
* diabetes complicated with coronary artery disease or vasculopathy
* alcoholism unweaned
* uncontrolled epilepsy and/or achievement of the central nervous system functions
* history of severe depressive syndrome
* presence or history of severe psychiatric condition, particularly severe depression, suicidal thoughts or attempted suicide
* decompensated liver cirrhosis
* severe myelosuppression
* psoriasis and sarcoidosis
* active disease condition or uncontrolled infection
* association with the yellow fever vaccine
* association with phenytoin in prophylaxis
* hypersensitivity against interferon or cyclophosphamide
* prior history of other malignancy except for: basal cell carcinoma of the skin, cervical intra-epithelial neoplasia and other cancer curatively treated with no evidence of disease for at least 3 years
* pregnancy, breast-feeding or absence of adequate contraception for fertile patients
* patients under guardianship, curatorship or under the protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-05-19 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
rate of patients with an immune response defined as "Tregs lymphocytes decrease ≥ 20% in blood by the flow cytometry technique" | at 3 months of the association CMC and Interferon-alpha

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Hôpital Nord Franche-Comté, Montbéliard